CLINICAL TRIAL: NCT02754921
Title: Percutaneous Dilatational Tracheostomy: Ultra-perc Single Stage Dilator Technique Versus Ciaglia Blue Dolphin Ballon Dilatation Technique for Intubated Unweanable ICU Patients
Brief Title: Percutaneous Dilatational Tracheostomy: Ultra-perc Versus Ciaglia Blue Dolphin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Sayed Mohamed Abbas (Other)
Responsible Party: Sponsor-Investigator, Mohamed Sayed Mohamed Abbas, Doctor, Al Mouwasat Hospital
Organization: Al Mouwasat Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSAT-2
Record Dates: First submitted 2016-04-25; First posted 2016-04-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: ICU Patients Dependant on Mechanical Ventilation : Safest Mode of Performing Percutaneous Tracheostomy Among ICU Ventilated Unweanable Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultra-perc (Experimental)
  Interventions: Procedure: percutaneous dilatational tracheostomy using Ultra-Perc
- Ciaglia Blue Dolphin (Experimental)
  Interventions: Procedure: Percutaneous dilatational tracheostomy using Ciaglia Blue Dolphin

INTERVENTIONS:
Procedure: percutaneous dilatational tracheostomy using Ultra-Perc — Procedure difficulties and complications faced while doing percutaneous dilatational tracheostomy using Ultra-Perc
  Arms: Ultra-perc
Procedure: Percutaneous dilatational tracheostomy using Ciaglia Blue Dolphin — Procedure difficulties and complications faced while doing percutaneous dilatational tracheostomy using Ciaglia Blue Dolphin
  Arms: Ciaglia Blue Dolphin

SUMMARY:
The aim of this study is to compare Ultra-perc single stage dilator technique with Ciaglia Blue Dolphin ballon dilatation technique for intubated unweanable ICU patients with respect to procedure difficulties and complications.

DETAILED DESCRIPTION:
The investigators conducted a prospective randomized trial to compare Ultra-perc single stage dilator technique (UP) and Ciaglia Blue Dolphin ballon dilatation technique (CBD) From January 2013 to December 2015.

The investigators compared the two groups as regards Procedure difficulties including difficult dilatation, difficult tube insertion, failed tube insertion, false passage and tracheal stoma over dilatation. and Procedure complications including cardiac arrest, pneumothorax, pneumomediastinum, subcutaneous emphysema, hemorrhage and lung atelectasis.

ELIGIBILITY:
Inclusion Criteria:

* sepsis
* cerebrovascular accidents
* cervical cord injury
* traumatic brain injury
* post arrest and chronic obstructive pulmonary disease

Exclusion Criteria:

* patient or family refusal
* emergency tracheostomy
* distorted abnormal anatomy
* bleeding diathesis
* morbid obesity
* previous tracheostomy
* infected surgical site
* Adult respiratory distress syndrome patients requiring high positive end expiratory pressure and high oxygen demands

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Procedure difficulties including difficult dilatation, difficult tube insertion, failed tube insertion, false passage and tracheal stoma over dilatation. | within 2 years
Procedure complications including cardiac arrest, pneumothorax, pneumomediastinum, subcutaneous emphysema, hemorrhage and lung atelectasis. | within 2 years

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Cianchi G, Zagli G, Bonizzoli M, Batacchi S, Cammelli R, Biondi S, Spina R, Peris A. Comparison between single-step and balloon dilatational tracheostomy in intensive care unit: a single-centre, randomized controlled study. Br J Anaesth. 2010 Jun;104(6):728-32. doi: 10.1093/bja/aeq087. Epub 2010 Apr 21. PMID 20413380